CLINICAL TRIAL: NCT05860842
Title: EXercise Capacity and TRAinability in Type 2 Diabetes (EXTRA-T2D)
Acronym: EXTRA-T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Università degli studi di Roma Foro Italico (Other)
Responsible Party: Principal Investigator, Giuseppe Pugliese, Professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-04
Record Dates: First submitted 2023-05-02; First posted 2023-05-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes; Exercise; Aging
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise training (Experimental): 6-month supervised exercise training program
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Six months of supervised combined exercise training program, consisting of 2 sessions/wk of 75 min each, followed by a six-month period of follow-up. Each session will comprise a 5-min warm-up, 30-min endurance exercise, 30-min resistance exercise, 5-min flexibility and 5-min cool-down.

SUMMARY:
Type 2 Diabetes (T2D) is a condition characterized by acelerated aging and is associated to multiple comorbidities, and physical fragility and disabilitiy, all of which reduce life expectancy and quality of life. Physical exercise has been demonstrated to have metabolic and cardiovascular benefits in T2D. Also, lack of exercise and sedentary behavior are major predictors of cardiovascular morbidity and mortality and all-cause mortality. Some evidence suggests that individuals with T2D have a reduced exercise capacity and exercise tollerance compared to non-diabetic individuals.The reasons behind such difference are not thoroughly explored, but may be connected to acute and chronic effects of hyperglycemia. Reduced trainability might be a marker of early aging and physical disalbility. This study aims to define respiratory, cardiovascular, neuromuscular, inflammatory, hormonal and metabolic determinants of trainability in persons with T2D. Results will help to answer the question whether it is the low trainability that reduces exercise capacity or it is the low exercise participation that determines a low exercise capacity.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is an age-related disease that is considered a condition of accelerated aging. It is in fact associated with multimorbidity, frailty and physically disability in older adults substantially impairing quality of life as well as with a reduced lifespan due to the occurrence of acute and, particularly, chronic complications, the most important of which is cardiovascular disease (CVD).

Reduced exercise capacity as a predictor of adverse outcomes in aging and age-related diseases. Physical inactivity and sedentary behavior have shown to be associated with increased all-cause and CVD morbidity and mortality in the general population and in people with diabetes. Both cardiorespiratory and muscle fitness have been shown to be independent predictors of death and to compensate for increased fatness, at least in part. In particular, exercise capacity or tolerance, i.e., the maximum amount of physical exertion that an individual can sustain, has been shown to predict mortality beyond traditional CVD risk factors and proposed as prognostic variable to be included in predictive algorithms in asymptomatic aging individuals or in those suffering from chronic disorders such as T2D. It can be assessed by cardiopulmonary exercise testing and usually measured as peak power output (PPO or peak work) or peak oxygen consumption (VO2peak). Though also dependent on the individual genetic background, the level of physical fitness/exercise capacity is largely determined by the amount of physical activity (PA), which is therefore strongly recommended in the general population and in people with T2D, together with reduction (and break) of sedentary time, which exerts detrimental effects independent of PA. In patients with T2D, in addition to providing overall health benefits, PA/exercise is effective in improving glucose control, CVD risk factors, and well-being, as also shown by our group.

Several studies have shown that patients with T2D have a reduced exercise capacity or tolerance as compared with non-diabetic individuals, though other reports failed to show any defect, especially if blood glucose is well-controlled. Studies investigating the mechanisms underlying the impaired exercise (aerobic) capacity have reported abnormalities in the ability of (a) lung to oxygenate arterial blood; (b) heart and vascular system to meet the circulatory demands; and (c) peripheral tissues to extract oxygen. In particular, decreased ventilatory efficiency, reduced peripheral oxygen extraction, impaired heart rate adjustment, and lower anaerobic threshold, have been shown in T2D individuals compared to non-diabetic subjects. In addition, T2D patients showed neuromuscular impairment with increased muscular fatigability. Our group has contributed to characterize the neuromuscular dysfunction of T2D by showing a reduction of isometric and dynamic muscle strength and endurance.

The reasons for the lower exercise capacity in the aging T2D population are unclear.

However, due to the cross-sectional design of most of the existing studies, the reasons for the lower exercise capacity in T2D patients are still unclear. On the one hand, these individuals might exercise less than non-diabetic individuals, as shown by several reports, consistent with the known role of physical inactivity and sedentary behavior as risk factors for the development of the disease. On the other hand, people with T2D might respond less to exercise training (reduced trainability), due to effects of hyperglycemia. These effects include the acute impact of poor glycemic control, with several deficits at least partially reversible upon improvement of HbA1c levels, and the chronic consequences of hyperglycemia, with subtle impairments in ventilatory, cardiorespiratory and neuromuscular function occurring prior to the onset of overt complications, the relation of which with reduced exercise capacity is well-established. In addition, a reduction in VO2 peak has been observed in first-degree relatives of T2D individuals versus accurately matched controls suggesting a possible role of the genetic background predisposing to T2D. Another mechanism which might be involved in the reduced exercise capacity and trainability is the chronic low-grade inflammation characterizing patients with T2D and the metabolic syndrome and potentially counteracted by engaging these individuals in exercise training programs, as shown by our group.

Impaired exercise capacity and reduced trainability can be considered early markers of aging, cardiometabolic disorders and physical disability. Assessing exercise capacity and its cardiorespiratory and neuromuscular determinants may therefore predict adverse outcomes, aid in designing and implementing personalized training interventions, and serve as a tool for evaluating the effect of therapeutic strategies in aging people and/or individuals with T2D.

2. AIMS

This project is aimed at assessing trainability of patients with T2D in order to clarify:

a. whether reduced exercise capacity is due to an impaired response (trainability) or a reduced adherence to training; b. which are the mechanisms involved and the respiratory, cardiovascular, neuromuscular, inflammatory, hormonal, and metabolic parameters predicting trainability.

3. DESIGN AND METHODS

3.1 Design This is a single-center, open-label, longitudinal intervention study comparing T2D versus non-diabetic individuals entitled "EXercise capacity and TRAinability in Type 2 Diabetes (EXTRA-T2D)".

Participants will be engaged in:

1. a 6-month supervised aerobic and strength training program, to assess response (and impact of glycemic control);
2. a 6-month post-training follow-up, to assess adherence (and possible impact of detraining).

Measurements will be performed at baseline (T0), at the end of the 6-month training (T1), and at the end of the 6-month post-training follow-up (T2).

At enrollment, participants will be given an accelerometer and an activity diary to monitor activities of daily life throughout the entire 12-months period. At each of these time points, participants will be given the questionnaires for the assessment of PA, barriers to exercise, health-related quality of life (QoL), and psychological well-being. They will be then evaluated for the study endpoints on four different days, on days 1-3 at the Exercise Physiology Laboratory of the University of Rome "Foro Italico" and on day 4 at Sant'Andrea University Hospital (University of Rome "La Sapienza").

On day 1, the accelerometer and questionnaires will be collected and participants will undergo assessment of anthropometric parameters and ventilatory and cardiorespiratory function at rest, followed by a ramp incremental cycling test until task failure in order to assess endurance exercise capacity as peak power output (PPO) and ventilatory and cardiorespiratory function in response to exercise.

On day 2, the ramp test will be repeated, as previously suggested, in order to partition within-participant day-to-day variability from the assessment of trainability.

On day 3, participants will perform neuromuscular tests. On day 4, participants will undergo routine biochemical testing and blood sample collection as well as cardiac and muscle magnetic resonance imaging (MRI) (at T0 and T1 only).

3.1.1. Participants This study will enroll 24 patients with T2D, 12 females and 12 males, and 24 age-and sex-matched non-diabetic volunteers serving as control group.

Absence of complications will be assessed based on normal ECG, carotid and lower limb Doppler ultrasound, fundus oculi, albuminuria, eGFR, vibration perception threshold as measured by a biothesiometer. Additional criteria for non-diabetic participants are absence of CVD and renal disease, as assessed based on normal ECG, carotid and lower limb Doppler ultrasound, albuminuria, and eGFR.

3.1.2. Recruitment Patients with T2D will be recruited at the outpatient Diabetes Clinic of Sant'Andrea University Hospital (University of Rome "La Sapienza"). Patients fulfilling the above criteria will be identified by the Diabetologist, asked to sign a statement of informed consent, and subjected to a cardiologic examination for cardiovascular evaluation, including a resting ECG and, based on clinical judgment, an echocardiogram and/or an ECG treadmill test, to obtain clearance for participation in the trial.

The non-diabetic volunteers will be recruited among non-diabetic patients attending the Endocrinology Unit of Sant'Andrea University Hospital and the University personnel at both the Sant'Andrea University Hospital (University of Rome "La Sapienza") and the University of Rome "Foro Italico".

3.1.3. Intervention Both T2D patients and non-diabetic controls will perform a 6-month supervised exercise training program at the gym facility of the Center for Sports and Physical Exercise Medicine of the Foundation of the University of Rome "Foro Italico", equipped with high-tech, new-concept machines donated by Technogym (Cesena, Italy) to the University of Rome "Foro Italico" as a result of joint application of the two units involved in this project to a call of the Italian Diabetes Society.

The program will consist of 2 sessions/wk of 75 min each, consisting of 5-min warm-up, 30-min endurance exercise, 30-min resistance exercise, 5-min flexibility and 5-min cool-down. The training load will be monitored with the CR-10 Rating of Perceived Exertion (RPE) scale and the NASA task load index scale during each training session.

The 30-min endurance exercise bout will be performed on a cycle ergometer (Excite Live Run, Technogym S.p.A.) recording power output, while also measuring respiratory frequency (fR) and HR with a wearable device (Howdy Senior, ComfTech, Monza, Italy) and RPE. The work rate will be initially set at 50% of the PPO at the incremental test aiming for an RPE of 5/10 at the end of the bout, hence allowing for within session adjustments in power output to reach this target. A submaximal incremental test will also be performed every month to adjust exercise intensity progression and assess changes in fR, HR or RPE. The starting power output will be set at 30 W and increased by 10W every min until reaching the 85% of the HR peak achieved in the experimental test.

The 30-min resistance exercise bout will consist of 8 to 10 exercises involving large muscle groups including the use of electronically controlled resistance training machine (Biostrength, Technogym), equipped with sensors allowing for real-time guidance of movement execution, measurement of maximal dynamic force (1-Repetition maximum, 1RM), and post-training extraction of raw mechanical data. At the beginning of the training program, participants will perform 3 sets of 12 repetitions at 60% of 1RM using the leg press, chest press and low row Biostrength line machines. The 1RM test on the three machines will be repeated every 2 wks to change the 60% target accordingly.

In diabetic participants, glycemic variations will be monitored before, during and after each training session, by means of a glucose meter, to decide whether patients are ready to perform the exercise session or need carbohydrate integration or treatment adjustment, to avoid adverse events during the session and the following 6-48 hours (e.g., hypoglycemic events).

3.1.4. Outcome measures The primary endpoint is change in endurance exercise capacity, i.e., PPO. Secondary endpoints include changes in ventilatory, cardiorespiratory and neuromuscular, and inflammatory parameters. Anthropometric, metabolic and (in males only) hormonal parameters, adherence and barriers to exercise, health-related QoL, and psychological well-being will be also assessed.

These outcomes will be assessed in the whole cohort, to evaluate overall trainability, in females versus males separately, to assess sex differences, and in each individual, to identify patients at risk.

3.2. Measurements 3.2.1. Primary endpoint Exercise capacity will be measured as the PPO achieved at the end of the ramp incremental test, registered to the nearest second. The test will be performed at the Exercise Physiology Laboratory of the University of Rome "Foro Italico" on an electromagnetically braked cycle ergometer (Lode Excalibur Sport, Groningen, the Netherlands). After 2 min of baseline pedaling at 20 W, the power output will be increased by 1 W/s (20 W/min) until task failure (i.e., the inability to maintain pedaling cadence at 70 rpm for more than 10 s). Participants will be asked to maintain this cadence throughout any ramp test to eliminate the potentially confounding effect of cadence on responses measured with a metabolic cart (Quark PFT, Cosmed, Rome, Italy). Trainability will be measured for single participants as the percentage difference from the average PPO of the incremental tests at T1 and the average PPO of the two incremental tests at T0 (ΔPPO). The ΔPPO of both T2D and control groups will then be calculated and compared by averaging ΔPPO of single participants in each group.

3.2.2. Secondary endpoints Ventilatory function

The following parameters will be measured at the end of the ramp incremental test performed at the Exercise Physiology Laboratory of the University of Rome "Foro Italico":

1. Respiratory frequency (fR);
2. Perceived exertion and dyspnea, assessed every min during the rampThe incremental test along with ventilatory variables;
3. Ventilatory efficiency, measured as the minute ventilation (V̇E) to carbon dioxide output slope obtained during incremental exercise;
4. Resting pulmonary diffusion capacity for carbon monoxide (DLCO) and related subcomponents (i.e., pulmonary capillary volume and alveolar capillary membrane diffusing capacity);
5. Forced vital capacity and pulmonary function (maximum ventilatory ventilation, pulmonary volumes, maximal inspiratory pressure and maximal expiratory);
6. Ventilatory flow morphology. Cardiorespiratory function

The following parameters will be measured at the end of the ramp incremental test performed at the Exercise Physiology Laboratory of the University of Rome "Foro Italico":

1. V̇O2peak;
2. Ventilatory thresholds (first and second);
3. Metabolic efficiency, as V̇O2-work rate slope;
4. HR and HR recovery (HRR), computed by subtracting the HR value at 1 min after test end from the HR peak during the test;
5. Oxygen pulse, as V̇O2/HR ratio;
6. Blood pressure, measured before, during and after incremental test with an automatic machine integrated with the metabolic cart;
7. HR variability (HRV), as an index of sympathetic and parasympathetic function. Neuromuscular function Participants will perform different neuromuscular tests at the Exercise Physiology Laboratory of the University of Rome "Foro Italico" to comprehensively evaluate the neuromuscular function of the knee extensors, while measuring force and HDsEMG activity of vastus lateralis (VL) and vastus medialis (VM) of the dominant limb. Tests of maximal isometric force, sustained contractions, trapezoidal changes in force and muscle endurance will be performed.

The following features will be extracted:

1. Muscle strength and endurance;
2. Neural drive;
3. Sources of neural drive;
4. Motor unit conduction velocity (MUCV);
5. Muscle fibre conduction velocity (MFCV);
6. Neuromuscular efficiency;
7. Neuromuscular manifestations of fatigue;
8. MU recruitment and derecruitment strategies;
9. Force steadiness. Cardiac and muscle MRI Cardiac and muscle MRI will be performed at the Radiology Unit of Sant'Andrea University Hospital (University of Rome "La Sapienza") in all participants at T0 and T1 only using a GE Signa 1.5 Tesla (GE Healthcare, Milan, Italy).

At cardiac MRI, left ventricular (LV) and right ventricular (RV) images will be obtained to obtain measures of:

1. LV and RV mass;
2. end-diastolic and end-systolic volumes;
3. stroke volumes;
4. ejection fraction;
5. cardiac output.

At thigh MRI, the following parameters wil be assessed:

1. muscle cross-sectional area;
2. intramuscular fat;
3. muscle density. Inflammatory profiling The following cytokines will be assayed in duplicate at the Department of Translational and Precision Medicine of the University of Rome "La Sapienza" by multiplex biometric ELISA-based immunoassay, using custom assay (Bioplex, Bio-Rad Lab) at T0, T1 and T2: Interleukin (IL)-1β, IL-2, IL-4, IL-6, IL-8, IL-12p70, interferon (IFN)-γ, and tumor necrosis factor (TNF)-α. Serum samples will be analyzed in the laboratory of the Principal Investigator.

Steroidomics Since aging and T2DM are associated with male hypogonadism and alteration of the hypothalamus-pituitary-adrenal axis, gonadal and adrenal steroids will be assayed in blood and salivary samples from male participants at T0, T1 and T2 at the Department of Experimental Medicine of the University of Rome "La Sapienza" using a recently validated in-house methodology capable of assessing up to 18 steroids simultaneously. Blood and salivary samples will be sent to Prof. Gianfrilli, Department of Experimental Medicine, Sapienza University of Rome, will be responsible for these analyses.

Metabolic parameters: Fasting glucose, insulin, triglycerides, total, HDL, and LDL cholesterol, and (in T2D patients only) HbA1c will be assessed at Laboratory Unit of Sant'Andrea University Hospital (University of Rome "La Sapienza") in all participants T0, T1 and T2.

Anthropometric parameters: Anthropometric characteristics (body weight and height with calculation of BMI, waist and hip circumference with calculation of waist-to-hip ratio, waist-to-height ratio, and A Body Shape Index [ABSI]) and body composition (by bioimpedance analysis) will be evaluated in all participants.

Exercise adherence and barriers: During the 12 months experimental period, each participant will be given a wrist-worn triaxial accelerometer (GENEActiv, Activinsights, Cambridgeshire, UK) and will also be requested to register daily activities by filling activity diaries. In addition, participants will be asked to complete the Italian version of the short form International Physical Activity Questionnaire. Perceived barriers to exercise will be also evaluated by using the Self-perceived Barriers for Physical Activity Questionnaire. Participants will be evaluated for health-related QoL and psychological well-being by the Italian version of the SF-36 Health Survey and the WHO-5 questionnaire, respectively.

3.3 STATISTICAL ANALYSIS

An a priori power analysis has been conducted for sample size estimation, using the G*power 3.1.9.2 Software. Given the paucity of studies reporting differences in trainability between T2D and healthy individuals, we have been cautious not to overestimate the effect size of any potential difference in PPO. Hence, a small effect size (i.e., 0.25) has been considered for the calculation, along with the following input information:

* Statistical test: ANOVA repeated measures, within-between interaction;
* α value: 0.05;
* 1-β: 0.8;
* Groups: 2;
* Measurements: 2;
* Correlation among repeated measures: 0.7. The resulting estimated sample size was 22 participants per group but, considering a dropping out of 10%, 24 participants per group will be recruited.

To assess differences in exercise capacity between T2D patients and non-diabetic controls, baseline (T0) values of the primary endpoint (PPO) and secondary endpoints (ventilatory, cardiorespiratory, and neuromuscular parameters) will be compared.

To assess differences in trainability between T2D patients and non-diabetic controls, change from baseline (T1-T0) in the primary endpoint and secondary endpoints will be compared.

To assess differences in adherence between T2D patients and non-diabetic controls, change from end-of-training (T2-T1) in the primary endpoint and secondary endpoints will be compared.

The unpaired Student's t test or the Mann-Whitney U test will be used for parametric and non-parametric variables, respectively.

In addition, univariate correlations by Spearman's rho and multivariable linear regression analyses will be used to identify correlates of change from baseline in exercise capacity (i.e., trainability).

ELIGIBILITY:
Inclusion Criteria:

* being below the recommended targets for MVPA and sedentary time (both healthy and diabetic individuals)

Additional inclusion criteria for participants with diabetes:

* HbA1c <7.5%
* dietary or pharmacological treatment excluding insulin
* disease duration >1 year
* free from chronic complications

Additional inclusion criteria for non-diabetic participants:

* absence of CVD and renal disease

Exclusion Criteria (both healthy and diabetic individuals):

* Smoking
* Any condition impairing ventilatory, cardiorespiratory and neuromuscular function, limiting or contraindicating PA, affecting conduct of the trial, reducing lifespan, and/or affecting the safety of intervention.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in peak power output (PPO) | 3 time points over 12 months: at baseline, after training (month 6) and after follow-up (month 12);
  Exercise capacity will be measured as the PPO achieved at the end of the ramp incremental test, registered to the nearest second. After 2 min of baseline pedaling at 20 W, the power output will be increased by 1 W/s (20 W/min) until task failure (i.e., the inability to maintain pedaling cadence at 70 rpm for more than 10 s). Participants will be asked to maintain this cadence throughout any ramp test to eliminate the potentially confounding effect of cadence on responses measured with a metabolic cart (Quark PFT, Cosmed, Rome, Italy). Trainability will be measured for single participants as the percentage difference from the average PPO of the incremental tests at T1 and the average PPO of the two incremental tests at T0 (ΔPPO). The ΔPPO of both T2D and control groups will then be calculated and compared by averaging ΔPPO of single participants in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pugliese, MD, PhD, Principal Investigator — University of Roma La Sapienza